CLINICAL TRIAL: NCT02859545
Title: Study to Understand Pain Experiences in Relationships
Acronym: SUPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Angelia Corley, Graduate Research Assistant, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ACorley
Record Dates: First submitted 2016-08-01; First posted 2016-08-09 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Chronic Pain
Keywords: chronic pain; pain; validation; couples; romantic relationships; emotional validation
MeSH Terms: conditions — Chronic Pain; Pain | interventions — Validation Studies as Topic; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Validation Training (Experimental): In this arm, the romantic partner of the individual with chronic pain receives training on how to validate which is provided by the research assistant.
  Interventions: Behavioral: Emotional Validation Training for Romantic Partners
- Education Training (Placebo Comparator): In this arm, the romantic partner of the individual with chronic pain receives training on how to ask questions about treatments, which is provided by the research assistant.
  Interventions: Behavioral: Chronic Pain Education Training for Romantic Partners

INTERVENTIONS:
Behavioral: Emotional Validation Training for Romantic Partners — In this intervention, romantic partners of individuals with chronic pain are trained individually by a research assistant. The romantic partner is trained on how to validate the individual with chronic pain's pain-related distress and given education about validation. This involves an approximately 45-minute brief, interactive training.
  Other Names: Validation
  Arms: Validation Training
Behavioral: Chronic Pain Education Training for Romantic Partners — In this intervention, romantic partners of individuals with chronic pain are trained individually by a research assistant. The romantic partner is trained on how to ask health professionals questions about treatment options and given health education about chronic pain. This involves an approximately 45-minute brief, interactive training.
  Other Names: Education
  Arms: Education Training

SUMMARY:
Chronic pain is a highly prevalent and costly health care problem. Yet, little is known about the optimal ways for health care providers and family members to respond to the distress expressed by people with chronic pain. The aim of the current study is to compare two models of responsiveness to identify responses that result in better functioning and adjustment. An experimental design will be used to test the extent to which emotional validation (e.g., an empathic response to distress) increases or decreases pain behaviors during physical activity. Romantic partners of individuals with chronic pain will be randomly assigned to receive validation or control training. Following training, people with chronic pain and their partners will engage in a discussion about pain and complete household tasks to examine the effects of partner training on communication, pain intensity, and pain behavior. Additionally, each individual in the couple will complete self-report measures after the discussion, after the household tasks, and one-month following the laboratory visit.

ELIGIBILITY:
Inclusion Criteria:

* Romantic couples who are married or living with each other for 6 months or longer or have been in a romantic relationship 2+ years.
* One individual in the couple must have chronic muscoskeletal pain, lasting 3 months or longer. Participants may have multiple pain sites.
* The individual with chronic pain must report that their pain occurs nearly daily.
* The individual with chronic pain must have an average pain intensity of 3 or greater on an 11-point scale (from 0: no pain to 10: worst pain imaginable)
* The individual with chronic pain must have an average pain interference of 3 or greater on an 11-point scale (from 0: does not interfere to 10: completely interferes)

Exclusion Criteria:

* One or both individuals in the couple are unable to speak, read, or write in English.
* Both individuals in the couple have chronic pain. Couples may consist of one individual with chronic pain and one individual with "minimal pain", which we define as having some aspects of chronic pain but not all (e.g., has had nearly daily pain for 4 months but rates their pain below 3 in regards to interference and intensity)
* One or both individuals in the couple have widespread pain (e.g., fibromyalgia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Pain Behavior (Behavioral coding) | During lab visit, during household tasks conducted in the laboratory, approx. 15 - 35 mins. after partner training (intervention)
  Pain behaviors (e.g., grimacing, guarding) measured with behavioral coding conducted by research assistants.
Pain Intensity (0 - 10 self-report rating scale) | During lab visit, during discussion task, approx. 5 minutes after partner training (intervention)
  The individual with chronic pain will be asked to report on the pain they experienced during the discussion with their partner, controlling for their baseline pain rating at the beginning of their laboratory visit.
Pain Intensity (0 - 10 self-report rating scale) | During lab visit, during household tasks, approx. 15 - 35 mins. after partner training (intervention)
  The individual with chronic pain will be asked to report on the pain they experienced during each household task (e.g., making a bed), controlling for baseline pain rating at the beginning of their laboratory visit.
Number of Partner Validating Responses (Behavioral coding) | During lab visit, during discussion task, approx. 5 minutes after partner training (intervention)
  Validating responses will be coded by research assistants.
Number of Partner Invalidating Responses (Behavioral coding) | During lab visit, during discussion task, approx. 5 minutes after partner training (intervention)
  Invalidating responses will be coded by research assistants.
Pain-Related Emotional Disclosures (Behavioral coding) | During lab visit, during household tasks, approx. 15 - 35 mins. after partner training (intervention)
  Behavioral coding by research assistants, accounting for activity level during household tasks.
Number of Partner Validating Responses (Behavioral coding) | During lab visit, during household tasks, approx. 15 - 35 mins. after partner training (intervention)
  Validating responses will be coded by research assistants
Number of Partner Invalidating Responses (Behavioral coding) | During lab visit, during household tasks, approx. 15 - 35 mins. after partner training (intervention)
  Invalidating responses will be coded by research assistants
Partner Instrumental support (Behavioral coding) | During lab visit, during household tasks, approx. 15 - 35 mins. after partner training (intervention)
  Partner instrumental support includes number of offers of assistance, acts of assistance, and behaviors that discourage physical activity, which will be measured by behavioral coding by research assistants
Individual with Chronic Pain Assistance Behavior (Behavioral coding) | During lab visit, during household tasks, approx. 15 - 35 mins. after partner training (intervention)
  Includes requests for assistance and accepting assistance, as measured by behavioral coding conducted by a research assistant

SECONDARY OUTCOMES:
Relationship Satisfaction (Questionnaire) | 1-month after the intervention
  Couples Satisfaction Index, Funk & Rogge, 2007. Both partners' self-reports of relationship satisfaction.
Interpersonal Closeness (Questionnaire) | During lab visit, during discussion task (approx. 5 mins. after intervention), and during household tasks (approx. 15 - 35 mins. after intervention), and 1-month after intervention
  Inclusion of Other in Self Scale, Aron, Aron, & Smollan, 1992. Both partners' self-reports of interpersonal closeness.
Perceived Partner Responsiveness (Questionnaire) | During lab visit, during discussion task (approx. 5 mins. after intervention), and during household tasks (approx. 15 - 35 mins. after intervention), and 1-month after intervention
  Reis et al., 2003.Both partners' self-reports on Perceived Partner Responsiveness.
Pain Intensity (Questionnaire) | 1-month after the intervention
  Brief Pain Inventory, Cleeland, 1992. The individual with chronic pain reports on their pain intensity using a 0 - 10 self-report scale, and indicates their average pain intensity over the last 24 hours.
Accuracy of Estimate of Individual with Chronic Pain's Pain Intensity | During lab visit, during discussion task (approx. 5 mins. after intervention), and during household tasks (approx. 15 - 35 mins. after intervention), and 1-month after intervention
  Romantic partner will be asked to estimate the individual with chronic pain's average pain intensity, which will be compared to the individual with chronic pain's report to assess accuracy.
Close other responses to pain and partner support (Questionnaire) | 1-month after the intervention
  West Haven-Yale Multidimensional Pain Inventory, Kerns, Turk, & Rudy, 1985. Both partners' reports of partner responses to pain and partner support, i.e., self-report for the partner, and other-report for the individual with chronic pain.
Perceived Partner Validation (Questionnaire) | During lab visit, during discussion task (approx. 5 mins. after intervention), and during household tasks (approx. 15 - 35 mins. after intervention), and 1-month after intervention
  Both partners' reports of partner's validation behavior, i.e., self-report for the partner, and other-report for the individual with chronic pain.
Perceived Partner Invalidation (Questionnaire) | During lab visit, during discussion task (approx. 5 mins. after intervention), and during household tasks (approx. 15 - 35 mins. after intervention), and 1-month after intervention
  Both partners report on partner's invalidation behavior, i.e., self-report for the partner, and other-report for the individual with chronic pain.
Ambivalence about emotional expression measured by Holding Back Scale (Questionnaire) | 1-month after the intervention
  * (Holding Back Scale; Pistrang & Barker, 1995)
  * (Holding Back Scale; Pistrang & Barker, 1995)
  * (Holding Back Scale; Pistrang & Barker, 1995)
  * (Holding Back Scale; Pistrang & Barker, 1995)
  * (Holding Back Scale; Pistrang & Barker, 1995) Holding Back Scale, Pistrang & Barker, 1995; Both partners report on individual with chronic pain's behavior.
Self- and Other-Oriented Distress (Questionnaire) | During lab visit, during discussion task (approx. 5 mins. after intervention) and during household tasks (approx. 15 - 35 mins. after intervention)
  Batson, Fultz, & Schoendrade, 1987. Both partners' self-report of self- and other-oriented distress.
Individual with Chronic Pain's Emotional Expression (Questionnaire) | During lab visit, during discussion task (approx. 5 mins. after intervention), and during household tasks (approx. 15 - 35 mins. after intervention), and 1-month after intervention
  Both partners' report on individual with chronic pain's emotional expression.
Individual with Chronic Pain's Pain Expression (Questionnaire) | During lab visit, during discussion task (approx. 5 mins. after intervention)and during household tasks (approx. 15 - 35 mins. after intervention)
  Both partners' report on individual with chronic pain's pain expression.
Perceived Division of Workload and Collaboration (Questionnaire) | After household tasks (approx. 35 - 45 mins. after intervention)
  Both partners' report on their perceptions of division of workload and collaboration during household tasks.
Satisfaction with the discussion (Questionnaire) | After discussion (approx. 15 mins. after intervention)
  Both partners' report on their satisfaction with the discussion.
Satisfaction with household tasks | After household tasks (approx. 35 - 45 mins. after intervention)
  Both partners' report

CONTACTS AND LOCATIONS:
Overall Officials: Angelia M Corley, M.A., Principal Investigator — Wayne State University
Locations (1):
- Wayne State University's Relationships and Health Lab, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No